CLINICAL TRIAL: NCT06960551
Title: Digital Transformation in Infertility Treatment: Effectiveness and Future Potential of a Comprehensive Mobile Web Application (Infertilitech)
Brief Title: Infertility Treatment
Acronym: ınfertilitech
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Simge Ozturk, Student, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Inonu5
Record Dates: First submitted 2025-04-03; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Infertility; Artificial Intelligence (AI)
Keywords: Obstetric Nursing; Primary Care Nursing; Infertility, Female; Web Browser
MeSH Terms: conditions — Infertility; Infertility, Female | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The project was planned as an experimental research with pretest-posttest experimental and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ınfertilitech group (Experimental): Before starting the project, the couples in the experimental group will be informed about the mobile application. The women will use the mobile application weekly for 3 months.
  4 times for at least 15 minutes each. To create motivation for use, women in the experimental group will be asked to motivational notification will be sent via the mobile application.
  Interventions: Other: ınfertility group
- control group (Other): Women in the control group will not receive any intervention. After collecting the post-test data in the project, the principle of benefit and equality Taking this into account, women and their husbands participating in the control group will be given the opportunity to use the mobile application free of charge for three months.
  Interventions: Other: control group

INTERVENTIONS:
Other: ınfertility group — Before starting the project, the couples in the experimental group will be informed about the mobile application. The women will use the mobile application weekly for 3 months.
  4 times for at least 15 minutes each. To create motivation for use, women in the experimental group will be asked to motivational notification will be sent via the mobile application.
  Arms: ınfertilitech group
Other: control group — Women in the control group will not receive any intervention. After collecting the post-test data in the project, the principle of benefit and equality Taking this into account, women and their husbands participating in the control group will be given the opportunity to use the mobile application free of charge for three months.
  Arms: control group

SUMMARY:
The primary objective of this project is to increase the treatment compliance and success of infertile couples based on the Knowledge-Motivation-Behavioral Skills model.

To develop a mobile web application and evaluate its effectiveness with scientific methods.

The secondary aim was to evaluate the effect of using a mobile application on Infertility Affect Status, Self-Efficacy, Infertility Adjustment and State-Trait Anxiety.

effect of the impact of the study.

DETAILED DESCRIPTION:
Infertility is a serious health problem affecting 8-12% of couples worldwide. This situation causes couples to face significant biopsychosocial and economic difficulties. Infertility process needs a multidisciplinary approach due to the diversity of etiological factors and complexity of treatment options. Especially in patriarchal societies, the problem of infertility may lead to negativities such as divorce, polygamy and social exclusion. In Turkey, the cultural importance of having children increases the psychological pressure on infertile couples. The coverage of infertility treatment by public institutions is limited. Therefore, couples often have to turn to the private sector and face high costs. Currently, infertile couples' sources of access to information are largely limited to the web pages of private infertility centres. In this context, the development of an evidence-based, reliable and free mobile web application for infertile couples emerges as a critical need. The main aim of this project is to develop a mobile web application to increase the treatment compliance and success of infertile couples and to evaluate its effectiveness with scientific methods. Original contributions are as follows:

* Creating a national comprehensive and culturally sensitive mobile web application different from the existing web pages on infertility. Regular updating and sharing of evidence-based medical and supportive treatment methods.
* Providing a structure that includes women as well as their husbands and family members in the process.

Inclusion of non-pharmacological methods (mindfulness etc.) in addition to medical treatments.

* Providing personalised information with the Ask Me module supported by artificial intelligence.
* R&D and scientific testing of the application with a randomised controlled trial.

In the second phase of the project, a randomised controlled study will be conducted with 74 individuals in the experimental group and 74 individuals in the control group who are treated in two infertility centres and who are determined by G-power. In the project, individuals in the experimental group will be asked to use the application for at least three months. Data will be collected using the Participant Information Form, measurement tools for infertility treatment compliance and success, and Mobile Application Evaluation Form. The user experience, interaction level and the effects of the application on increasing adherence to treatment will also be analysed. With the successful completion of the project, it is envisaged that a national mobile application will be created, the application will be translated into different languages to expand its usage area and economic sustainability will be ensured. In addition, it is planned to contribute to health policies in line with the scientific data obtained, to increase the effectiveness of digital health solutions for infertility and to facilitate access to health services.

ELIGIBILITY:
Inclusion Criteria:

for women;

* To be between the ages of 18-45,
* Being diagnosed with primary infertility,
* To be able to read, write and understand Turkish,
* Not having a disability to use a smartphone,
* Being at the stage of agreeing to start infertility treatment (initial period of treatment),
* Using the mobile app at least 4 times a week for 15 minutes each for 3 months for partner
* Volunteer to participate in the project,
* Not having a disability to use a smartphone,
* Using the mobile app at least 1 time/15 minutes per week for 3 months

Exclusion Criteria:

for women

* Incomplete answers to forms,
* Not using the mobile app at all for a week,
* Wanting to leave the study,
* Voluntary discontinuation of infertility treatment for partner
* Incomplete completion of the forms (uMARS and State-Trait Anxiety Inventory),
* Not using the mobile app at all for two weeks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Infertility Adjustment Scale | three months
  The Turkish validity and reliability of the scale developed by Glover et al. was analyzed by Arslan Özkan et al. was conducted. The scale is six-point Likert-type and consists of 12 items. The scale is only administered to women. Scores that can be obtained from the scale are 12-72 ranges between the two scales. Increasing scores on the scale indicate an increase in maladjustment to loss of fertility. Cronbach's alpha coefficient was determined as 0.77

SECONDARY OUTCOMES:
Infertility Affect Scale | three months
  The scale developed by Akyüz et al. (2008) assesses women's level of being psychologically affected by infertility. determines. The scale is four-point Likert-type and consists of 21 items. There are 16 positive and 5 negative items in the scale. The items in the scale Items 3, 10, 13, 14 and 21 are expressed negatively and these items are reverse coded. Scores that can be obtained from the scale range between 21-84 varies. The higher the scores obtained from the scale, the higher the level of psychological impact of infertility. Cronbach alpha coefficient was determined as 0.93
Participant Information Form | three months
  The participant information form developed by the researchers in line with the literature consists of two parts. Form one age, educational status, occupation, income, duration of marriage, duration of infertility, and knowledge of the cause of infertility, cause of infertility, diagnosed infertility, frequency of past infertility treatment, name of past infertility treatment, current the infertility treatment received, the planned stage of infertility treatment, the medication currently being taken, any incorrect or faulty medication used during treatment practice status, use of traditional methods for infertility treatment, traditional methods used, 18 questions including traditional methods used takes
Infertility Self-Efficacy Scale-Short Form | three months
  The Turkish validity and reliability of the scale developed by Cousineau et al. Özkan et al. (2012). The scale is applied only to women. The scale is four-point Likert-type and consists of 8 items. In the scale All items are positive and the scores that can be obtained from the scale vary between 8-32. As the scores obtained from the scale increase, individuals' self-efficacy perception increased. Croncah alpha coefficient of the scale was determined as 0.78
State-Trait Anxiety Inventory | three months
  The Turkish validity and reliability of the inventory developed by Spielberger et al. Compte (1983). The four-point Likert-type inventory, which is suitable for both women and men, consists of 40 items. It consists of two subscales, state and trait anxiety. The State Anxiety Scale assesses how the individual feels at a certain moment and under certain conditions. It evaluates their feelings about the situation they are in by describing how they feel. The Trait Anxiety Scale assesses how the individual usually feeling of being a victim. Both scales consisted of twenty items each. The total score value obtained from the scale ranges between 20 and 80. It was determined that as the score increased, the level of anxiety increased and as the score decreased, the level of anxiety decreased.
User Version of the Mobile Application Rating Scale | three months
  Calik et al. (2022) conducted the Turkish validity and reliability study of the scale developed by Calik et al. Quality of health practices uMARS, developed to assess quality, consists of five subscales, a five-point Likert-type scale and 20 items. Four subscales are objective and quality rating. These are participation (5 items), functionality (4 items), aesthetics (3 items) and knowledge (4 items). One subscale is evaluated subjectively (4 items). The perceived impact subscale has 6 items and evaluates the impact of the perception of the application by the user. A minimum of 20 and a maximum of 100 points are obtained from the scale. The higher the score, the higher the validity of the mobile application. The project, the application password is available for women as well as their spouses. will be given. In the project, the UMARS form will be used in the post-test to assess the spouses' satisfaction with the mobile application/WhatsApp. will be asked to fill in the form.

CONTACTS AND LOCATIONS:
Overall Officials: Simge Öztürk, Ph.D, Principal Investigator — Inonu University

IPD SHARING:
Plan to Share IPD: No